CLINICAL TRIAL: NCT06761053
Title: Can the Albumin/High Sensitive C-reactive Protein Ratio be Utilized for Predicting Gestational Diabetes Mellitus Diagnosis or the Adverse Outcomes
Brief Title: Can Albumin/C-reactive Protein Ratio be Utilized for Predicting Gestational Diabetes Diagnosis or the Adverse Outcomes
Acronym: Alb/hsCRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ALI BAHADIRLI (Other)
Collaborators: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Sponsor-Investigator, ALI BAHADIRLI, M.D., Mustafa Kemalpasa Government Hospital
Organization: Mustafa Kemalpasa Government Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-KAEK-25
Record Dates: First submitted 2024-12-28; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: Gestational diabetes mellitus; Albumin; C-reactive protein; Pregnancy complications; Clinical marker
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: All participants underwent the same screening and diagnostic protocol (GCT and possibly OGTT) to assess glucose tolerance or diagnose gestational diabetes mellitus (GDM). They were not divided into separate groups to receive distinct interventions or different sequences of the same intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GDM Group (Experimental Arm) (Experimental): This arm included 46 participants diagnosed with GDM following the 100-gram oral glucose tolerance test (OGTT) and meeting the Carpenter and Coustan diagnostic criteria for GDM. These participants showed higher levels of fasting glucose and C-reactive protein (CRP), and a higher hsCRP/albumin ratio compared to the control group. The study aimed to explore the relationship between the albumin/hsCRP ratio and GDM, along with the associated pregnancy complications and perinatal outcomes.
  Interventions: Diagnostic Test: Intervention/Exposure for the GDM Group (Experimental Arm)
- Control Group (Control Arm) (Other): This arm consisted of 100 participants who had normal glucose tolerance, identified through the glucose challenge test (GCT) with results below 140 mg/dL, and did not meet the criteria for GDM on the OGTT. The control group was used for comparison to assess the differences in albumin/hsCRP ratios, glucose levels, and pregnancy outcomes between women without GDM and those diagnosed with GDM.
  Interventions: Diagnostic Test: Intervention/Exposure for the Control Group

INTERVENTIONS:
Diagnostic Test: Intervention/Exposure for the GDM Group (Experimental Arm) — Gestational Diabetes Diagnosis: The intervention for this group involves the diagnostic procedure of the 100-gram oral glucose tolerance test (OGTT) after an initial glucose challenge test (GCT) with a result equal to or greater than 140 mg/dL. The test assesses fasting plasma glucose and post-glucose consumption plasma glucose levels at 1 hour and 2 hours, which is used to diagnose GDM.
  Biomarker Analysis: The albumin to high-sensitivity C-reactive protein (hsCRP) ratio is measured as a biomarker to explore its potential role in GDM diagnosis and related pregnancy outcomes.
  Arms: GDM Group (Experimental Arm)
Diagnostic Test: Intervention/Exposure for the Control Group — Glucose Challenge Test (GCT): The control group participants are exposed to the glucose challenge test (GCT), where plasma glucose levels are measured one hour after the consumption of 50 grams of glucose. If their glucose levels are below 140 mg/dL, they are categorized as not having GDM.
  Biomarker Analysis: Similar to the GDM group, the albumin to hsCRP ratio is measured for participants in the control group to compare the biomarker levels between those with and without GDM.
  Arms: Control Group (Control Arm)

SUMMARY:
This study provides a comprehensive evaluation of the potential utility of the albumin/high-sensitivity C-reactive protein (hsCRP) ratio in diagnosing gestational diabetes mellitus (GDM) and predicting adverse pregnancy outcomes. The findings underscore the role of systemic inflammation, represented by hsCRP levels, in GDM's pathophysiology and associated complications.

The results align with existing literature linking inflammation markers, such as hsCRP, to GDM and other metabolic disturbances during pregnancy. The significant differences in hsCRP and albumin/hsCRP ratios between the GDM and control groups reinforce the importance of these markers in identifying at-risk pregnancies. Moreover, the ROC analysis, with a statistically significant AUC, highlights the predictive capability of these ratios, suggesting their incorporation into clinical practice could improve early identification and management of GDM.

The discussion further situates these findings within a broader context of research, emphasizing the inflammatory origins of GDM and their implications for maternal and neonatal health. Future research could explore the integration of inflammatory markers with other diagnostic tools to enhance the sensitivity and specificity of GDM screening protocols. This approach may ultimately contribute to reducing the burden of GDM-related complications and improving pregnancy outcomes.

DETAILED DESCRIPTION:
Introduction

Pregnancy necessitates a fine balance between pro- and anti-inflammatory processes to establish a favorable uterine environment. Disruptions in this balance, such as inflammation, are associated with adverse outcomes, including gestational diabetes mellitus (GDM). GDM prevalence varies globally, influenced by ethnicity, diagnostic criteria, and cultural differences, ranging from 1% to 28%. In Europe, the prevalence is approximately 5-10%, posing significant risks for maternal and neonatal health. Universal screening between 24-28 weeks of gestation is widely recommended.

Primary GDM risk factors include advanced maternal age, obesity, and inflammation. Adipose tissue, an endocrine organ, secretes adipokines such as leptin and adiponectin, which impact glucose metabolism, particularly in obesity-related insulin resistance. Pregnancy-induced insulin resistance ensures fetal glucose supply, but insufficient pancreatic beta-cell compensation may lead to GDM. These mechanisms underscore the rationale for mid-gestation GDM screening.

Although glucose tolerance tests are considered safe, concerns about glucose ingestion during pregnancy highlight the need for innovative diagnostic approaches. Given GDM's inflammatory underpinnings, markers of acute inflammation could enhance diagnostic accuracy. This study evaluates the albumin/high-sensitivity C-reactive protein (hsCRP) ratio's utility in diagnosing GDM and predicting adverse outcomes.

Material and Methods

Study Design and Participants

This prospective clinical cohort study was conducted at a training and research hospital with ethics committee approval. Pregnant women at 24-28 weeks of gestation, determined by last menstrual period and first-trimester ultrasonography, were enrolled. The study adhered to the Declaration of Helsinki principles, with participants providing written informed consent for data collection and analysis.

GDM Screening and Diagnosis

The glucose challenge test (GCT) measured plasma glucose one hour after consuming 50 grams of glucose. Participants with GCT results ≥140 mg/dL underwent a 100-gram oral glucose tolerance test (OGTT) after a standardized three-day diet. OGTT diagnostic criteria included fasting plasma glucose (FPG) levels and glucose measurements at 1-hour and 2-hour intervals post-glucose ingestion, categorized per Carpenter and Coustan criteria. Some participants underwent 75-gram OGTT, with diagnostic thresholds similarly defined.

Laboratory Measurements

Blood samples were analyzed in the hospital laboratory. Albumin levels were measured using the bromocresol green method, and hsCRP levels were assessed using nephelometry. The albumin/hsCRP ratio was calculated accordingly.

Exclusion Criteria

Participants with pre-gestational diabetes, BMI >30, age >35, GDM history, macrosomic delivery history, unexplained fetal loss, type II diabetes family history, endocrinology diseases, liver or renal disease, or systemic/local infection were excluded.

Data Collection and Review

Antenatal visit records and delivery outcomes were reviewed for complications, including preeclampsia, gestational hypertension, amniotic fluid abnormalities, fetal anomalies, preterm labor, and postpartum hemorrhage. Neonatal outcomes, such as birth weight, APGAR scores, NICU admission, and stillbirth, were also assessed.

Statistical Analysis

The Shapiro-Wilk test assessed variable normality. Normally distributed variables were compared using Student's t-tests; non-normally distributed variables were analyzed with Mann-Whitney U tests. Categorical variables were compared using Chi-square or Fisher's exact tests. ROC curve analysis evaluated the albumin/hsCRP ratio's predictive potential, reporting AUC, sensitivity, specificity, and cut-off values. Analyses were performed using SPSS 22 and MedCalc 19.5.6, with p<0.05 considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 24 and 28 weeks of gestation.
* Gestational age confirmed by both last menstrual period and first-trimester ultrasonography.
* Signed informed consent for data collection, analysis, and use for research.

Exclusion Criteria:

* Pre-gestational diabetes mellitus.
* BMI > 30.
* Age > 35 years.
* A history of gestational diabetes mellitus (GDM).
* Previous delivery of macrosomic infants.
* Unexplained fetal loss.
* Family history of type II diabetes mellitus.
* Any endocrinological disease.
* Liver disease, renal disease, or other significant systemic or local infections.

Max Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 146 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-07-03 (Actual)

PRIMARY OUTCOMES:
Comparison of Albumin to High-Sensitivity C-Reactive Protein (hsCRP) Ratio Between GDM and Control Groups | At the time of GDM diagnosis (during the 24-28 weeks of gestation) and at the end of the study.
  This primary outcome measure assesses the difference in the albumin to hsCRP ratio between pregnant women diagnosed with gestational diabetes mellitus (GDM) and those in the control group with normal glucose tolerance. The albumin/hsCRP ratio is explored as a potential biomarker for GDM diagnosis and its relationship with pregnancy-related outcomes.

SECONDARY OUTCOMES:
Prevalence of Pregnancy Complications in Women with GDM vs. Control Group | During pregnancy and up to delivery (final pregnancy outcome assessment).
  This outcome measure evaluates the occurrence of pregnancy complications, including threatened labor, preeclampsia, acute fetal distress, and other related conditions in women diagnosed with GDM compared to the control group.
Gestational Age at Delivery in GDM vs. Control Group | At the time of delivery.
  This outcome measure examines the difference in gestational age at delivery between the two groups. The study aims to assess whether GDM affects the timing of delivery.
Birth Weight and Neonatal Outcomes in GDM vs. Control Group | At birth (within 24 hours after delivery).
  This measure compares the birth weight, APGAR scores, and neonatal intensive care unit (NICU) admission rates between women diagnosed with GDM and the control group.
Change in Plasma Glucose Levels from GCT to OGTT in GDM and Control Groups | During the 24-28 weeks of gestation (at the time of GCT and OGTT).
  This outcome measures the change in plasma glucose levels after the GCT and the subsequent 100-gram oral glucose tolerance test (OGTT) in both groups, assessing glucose tolerance and its relationship with GDM.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Bahadirli, M.D., Principal Investigator — Bursa City Hospital
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, University of Health Sciences, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
As per the facility's policy, individual participant data (IPD) will not be shared. The facility does not currently permit the sharing of such data for research purposes. We appreciate your understanding and respect for this policy.

REFERENCES:
- [Background] Eckart A, Struja T, Kutz A, Baumgartner A, Baumgartner T, Zurfluh S, Neeser O, Huber A, Stanga Z, Mueller B, Schuetz P. Relationship of Nutritional Status, Inflammation, and Serum Albumin Levels During Acute Illness: A Prospective Study. Am J Med. 2020 Jun;133(6):713-722.e7. doi: 10.1016/j.amjmed.2019.10.031. Epub 2019 Nov 18. PMID 31751531
- [Background] Levitt DG, Levitt MD. Human serum albumin homeostasis: a new look at the roles of synthesis, catabolism, renal and gastrointestinal excretion, and the clinical value of serum albumin measurements. Int J Gen Med. 2016 Jul 15;9:229-55. doi: 10.2147/IJGM.S102819. eCollection 2016. PMID 27486341
- [Background] Keenan-Devlin LS, Caplan M, Freedman A, Kuchta K, Grobman W, Buss C, Adam EK, Entringer S, Miller GE, Borders AEB. Using principal component analysis to examine associations of early pregnancy inflammatory biomarker profiles and adverse birth outcomes. Am J Reprod Immunol. 2021 Dec;86(6):e13497. doi: 10.1111/aji.13497. Epub 2021 Sep 19. PMID 34477256
- [Background] Amirian A, Rahnemaei FA, Abdi F. Role of C-reactive Protein(CRP) or high-sensitivity CRP in predicting gestational diabetes Mellitus:Systematic review. Diabetes Metab Syndr. 2020 May-Jun;14(3):229-236. doi: 10.1016/j.dsx.2020.02.004. Epub 2020 Mar 16. PMID 32247209
- [Background] Sifnaios E, Mastorakos G, Psarra K, Panagopoulos ND, Panoulis K, Vitoratos N, Rizos D, Creatsas G. Gestational Diabetes and T-cell (Th1/Th2/Th17/Treg) Immune Profile. In Vivo. 2019 Jan-Feb;33(1):31-40. doi: 10.21873/invivo.11435. PMID 30587599
- [Background] Liu W, Huang Z, Tang S, Zhang Z, Yu Q, He J. Changes of Serum Sex Hormone-Binding Globulin, Homocysteine, and Hypersensitive CRP Levels during Pregnancy and Their Relationship with Gestational Diabetes Mellitus. Gynecol Obstet Invest. 2021;86(1-2):193-199. doi: 10.1159/000515085. Epub 2021 Apr 27. PMID 33906193
- [Background] Bo S, Signorile A, Menato G, Gambino R, Bardelli C, Gallo ML, Cassader M, Massobrio M, Pagano GF. C-reactive protein and tumor necrosis factor-alpha in gestational hyperglycemia. J Endocrinol Invest. 2005 Oct;28(9):779-86. doi: 10.1007/BF03347566. PMID 16370555
- [Background] Maged AM, Moety GA, Mostafa WA, Hamed DA. Comparative study between different biomarkers for early prediction of gestational diabetes mellitus. J Matern Fetal Neonatal Med. 2014 Jul;27(11):1108-12. doi: 10.3109/14767058.2013.850489. Epub 2013 Oct 22. PMID 24090161
- [Background] Eades CE, Cameron DM, Evans JMM. Prevalence of gestational diabetes mellitus in Europe: A meta-analysis. Diabetes Res Clin Pract. 2017 Jul;129:173-181. doi: 10.1016/j.diabres.2017.03.030. Epub 2017 May 9. PMID 28531829
- [Background] Saeedi M, Cao Y, Fadl H, Gustafson H, Simmons D. Increasing prevalence of gestational diabetes mellitus when implementing the IADPSG criteria: A systematic review and meta-analysis. Diabetes Res Clin Pract. 2021 Feb;172:108642. doi: 10.1016/j.diabres.2020.108642. Epub 2021 Jan 13. PMID 33359574
- [Background] Sharma AK, Singh S, Singh H, Mahajan D, Kolli P, Mandadapu G, Kumar B, Kumar D, Kumar S, Jena MK. Deep Insight of the Pathophysiology of Gestational Diabetes Mellitus. Cells. 2022 Aug 28;11(17):2672. doi: 10.3390/cells11172672. PMID 36078079